CLINICAL TRIAL: NCT07316894
Title: International Delphi Consensus on the Universal Definition and Diagnosis of Iatrogenic Withdrawal Syndrome in Adult ICU Patients
Brief Title: IWS Diagnosis Criteria Consensus
Status: Recruiting | Type: Observational
Sponsor: ELIAS Emergency University Hospital (Other)
Collaborators: University of Rome Tor Vergata (Other); Boston University (Other); Carol Davila University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Emanuel Moisa, MD, PhD, DESAIC, Assistant Professor and Specialist of Anaesthesia and Critical Care Medicine,, ELIAS Emergency University Hospital
Other Study IDs: 10122025
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Iatrogenic Withdrawal Syndrome
Keywords: iatrogenicwithdrawalsyndrome; ICU; delphiconsensus
MeSH Terms: interventions — Intensive Care Units; Anesthesia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ICU, Anesthesiology and Psychiatry specialists consensus on the diagnosis of IWS. — This is a new and originally developed questionnaire comprising of 19 questions. Out of 19 questions, 17 use a 7-point Likert scale response, one uses a Yes/No type of answer and one has open answers.

SUMMARY:
This is an International Delphi Consensus on the Definition and Diagnosis of Iatrogenic Withdrawal Syndrome in adult critically ill patients. It involves the anonymous completion of a questionnaire using a 7-point Likert scale.

ELIGIBILITY:
Inclusion Criteria:

* At least 5 years of experience or training or research in the field of Intensive Care Medicine, Anesthesiology or Psychiatry

Exclusion Criteria:

* Not a specialist in the fields of Intensive Care Medicine, Anesthesiology or Psychiatry

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Professionals from the following medical specialties are eligible: Intensive Care Medicine, Anesthesiology or Psychiatry.
  Participants to this Delphi Consensus must have at least 5 years of experience in their field.
  Academic title or previous research published in the field of Iatrogenic Withdrawal Syndrome are not mandatory.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-12-13 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Criteria of IWS | 4 monts
  The diagnostic criteria of IWS will be determined based on the items reaching the consensus

CONTACTS AND LOCATIONS:
Overall Officials: Emanuel Moisa, Assist. Prof., MD, PhD, DESAIC, Principal Investigator — Elias Emergency University Hospital of Bucharest, Carol Davila University of Medicine and Pharmacy, Bucharest; Federico Bilotta, Professor, MD, PhD, Study Chair — Tor Vergata University of Rome
Locations (1):
- Elias Emergency University Hospital, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: Yes
The exact number of answers provided for each question from the questionnaire will be provided, as well as all the Delphi rounds in which agreement was or was not met.
  Demographic data about experts in order to ensure their eligibility.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Moisa E, Tuculeanu G, Corneci D, Negoita SI, Bilotta F. Iatrogenic withdrawal syndrome in adult intensive care unit: a scoping review. Front Med (Lausanne). 2025 Jul 23;12:1573363. doi: 10.3389/fmed.2025.1573363. eCollection 2025. PMID 40771468